CLINICAL TRIAL: NCT02796092
Title: Fibered Platinum Coils vs Vascular Plugs in Pelvic Varices Embolization for the Treatment of Pelvic Congestion Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Group of Research in Minimally Invasive Techniques (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GTM-01
Record Dates: First submitted 2016-05-27; First posted 2016-06-10 (Estimated); Results first posted 2016-10-26 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2017-02

CONDITIONS: Pelvic Congestion Syndrome
Keywords: Pelvic Congestion Syndrome; Pelvic Venous Insufficiency; Chronic pelvic pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fibered platinum coils (Active Comparator): Embolization of the pelvic veins with platinum fibered coils (Nester. Cook Europe, Bjaeverskov, Denmark)
  Interventions: Device: Fibered platinum coils
- Vascular plugs (Experimental): Embolization of the pelvic veins with vascular plugs (Amplatzer Vascular Plugs II. St. Jude Medical. St. Paul, MN, USA)
  Interventions: Device: Vascular plugs

INTERVENTIONS:
Device: Fibered platinum coils
  Other Names: Nester coils
  Arms: Fibered platinum coils
Device: Vascular plugs
  Other Names: Amplatzer vascular plugs
  Arms: Vascular plugs

SUMMARY:
This prospective randomized study compares the safety and efficacy of two different embolizing agents for the treatment of pelvic congestion syndrome: fibered platinum coils and vascular plugs.

DETAILED DESCRIPTION:
This prospective randomized study compares the safety and efficacy of two embolizing agents for the treatment of pelvic congestion syndrome: fibered platinum coils (Nester coils; Cook Medical) and vascular plugs (Amplatzer vascular plugs II; St. Jude Medical).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Presence of chronic abdominal or pelvic pain for more than 6 months
* >6 mm pelvic venous caliber measured by transvaginal US
* Presence of venous reflux OR presence of communicating veins assessed by transvaginal Doppler US

Exclusion Criteria:

* Diagnosed gynecological or pelvic pathology: endometriosis, pelvic inflammatory disease, postoperative adhesions, adenomyosis or leiomyoma
* Glomerular filtration rate <60 ml/min
* History of contrast reaction
* Patients not able to be followed up for at least one year

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-02; Primary Completion 2015-02 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Miguel A De Gregorio, MD, PhD, Principal Investigator — Universidad de Zaragoza
Locations (1):
- Lozano Blesa University Hospital, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited based on physician referral in a single specialized center between January 2014 and January 2015. The 1 year follow-up period was finished in February 2016.
Groups:
- Fibered Platinum Coils: Embolization of the pelvic veins with platinum fibered coils (Nester. Cook Europe, Bjaeverskov, Denmark)
  Fibered platinum coils
- Vascular Plugs: Embolization of the pelvic veins with vascular plugs (Amplatzer Vascular Plugs II. St. Jude Medical. St. Paul, MN, USA)
  Vascular plugs
Period: Overall Study
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Started | 50 | 50
Completed | 50 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All the patients were women referred from a vascular surgeon, diagnosed of pelvic congestion syndrome and pelvic varices by transvaginal ultrasound Doppler aged over 18.
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibered Platinum Coils | Vascular Plugs | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.00 (6.26) | 44.34 (8.45) | 42.67 (7.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 50 | 100
  Male | 0 | 0 | 0
Living children [Mean (Standard Deviation); unit: Children] | 1.86 (0.96) | 1.78 (0.71) | 1.82 (0.8)
Pre-treatment Visual Analogue Score [Mean (Standard Deviation); unit: units on a scale] — VAS is a subjective pain scale, scored from 1 to 10 (1 no pain; 10 worst pain possible)
  units on a scale | 7.14 (1.55) | 7.88 (1.01) | 7.51 (1.36)
Pain in orthostatic position [Number; unit: participants]
  YES | 48 | 50 | 98
  NO | 2 | 0 | 2
Pain in supine position [Number; unit: participants]
  YES | 7 | 6 | 13
  NO | 43 | 44 | 87
Dyspareunia [Number; unit: participants]
  YES | 27 | 27 | 54
  NO | 23 | 23 | 46
Dysmenorrhea [Number; unit: participants]
  YES | 27 | 35 | 62
  NO | 23 | 15 | 38
Urinary urgency [Number; unit: participants]
  YES | 7 | 6 | 13
  NO | 43 | 44 | 87
History of ovarian cystic disease [Number; unit: participants]
  YES | 22 | 21 | 43
  NO | 28 | 29 | 57
History of vaginal varicosities [Number; unit: participants]
  YES | 10 | 8 | 18
  NO | 40 | 42 | 82
History of vulvar varicosities [Number; unit: participants]
  YES | 18 | 19 | 37
  NO | 32 | 31 | 63
History of lower limb varices [Number; unit: participants]
  YES | 45 | 44 | 89
  NO | 5 | 6 | 11
History of lower limb varices surgery [Number; unit: participants]
  YES | 10 | 10 | 20
  NO | 40 | 40 | 80
Maximum right pelvic venous caliber [Mean (Standard Deviation); unit: mm] | 7.38 (1.19) | 7.36 (1.22) | 7.37 (1.20)
Maximum left pelvic venous caliber [Mean (Standard Deviation); unit: mm] | 6.78 (1.96) | 6.66 (1.55) | 6.72 (1.76)
Varicocele [Number; unit: participants]
  YES | 41 | 45 | 86
  NO | 9 | 5 | 14
Ovarian vein reflux [Number; unit: participants]
  YES | 40 | 35 | 75
  NO | 10 | 15 | 25
Waveform change in Valsalva's maneuver [Number; unit: participants]
  YES | 25 | 30 | 55
  NO | 25 | 20 | 45

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Scale
Description: Reduction of 4 points or more between subjective pain assessed by VAS prior to procedure (-4, -5,- 6, -7,-8,-9).
  VAS= visual analogue scale: it is a subjective pain scale, scored from 1 to 10 (1 no pain; 10 worst pain possible)
Time Frame: 12 months
Population: Population presenting pre-treatment pain (more than 1 in VAS)
Measure: Number; unit: participants
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 49 | 50
participants
  IMPROVEMENT | 47 | 48
  NO IMPROVEMENT | 2 | 2
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Assuming that both methods were equally effective, we did not use this primary outcome to calculate sample size. It was determined using our own retrospective data of patients from the year 2013, comparing the means of the procedure total time with both methods (41.20±4.66 vs 34.99±4.43 minutes). Ten patients in each group were considered enough to detect the above-mentioned differences with a α-error of 0.05 and 80% power, using a two-sided test; Test type: Superiority or Other; p > 0.999, Fisher Exact

2. Secondary Outcome: Improvement of Dyspareunia
Description: Disappearance or improvement of dyspareunia assessed by direct questioning before the procedure and 12 months after the procedure (YES/NO)
Time Frame: 12 months
Population: Population presenting pre-treatment dyspareunia
Measure: Number; unit: participants
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 27 | 27
participants
  IMPROVEMENT | 24 | 21
  NO IMPROVEMENT | 3 | 6
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p = 0.3, Fisher Exact

3. Secondary Outcome: Improvement of Urinary Urgency
Description: Disappearance or improvement of urinary urgency assessed by direct questioning before the procedure and 12 months after the procedure (YES/NO)
Time Frame: 12 months
Population: Population presenting pre-treatment urinary urgency
Measure: Number; unit: participants
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 7 | 6
participants
  IMPROVEMENT | 6 | 6
  NO IMPROVEMENT | 1 | 0
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p > 0.999, Fisher Exact

4. Secondary Outcome: Improvement of Dysmenorrhea
Description: Disappearance or improvement of dysmenorrhea assessed by direct questioning before the procedure and 12 months after the procedure (YES/NO)
Time Frame: 12 months
Population: Population presenting pre-treatment dysmenorrhea
Measure: Number; unit: participants
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 27 | 35
participants
  IMPROVEMENT | 24 | 31
  NO IMPROVEMENT | 3 | 4
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p > 0.999, Fisher Exact

5. Secondary Outcome: Satisfaction With the Procedure
Description: Overall satisfaction with the procedure via telephone survey (scaled from 0 to 9).
  Patients answered just one question. Are you satisfied with the procedure? Being 0 = Completely unsatisfied, I regret having undergone a embolization procedure 9=Totally satisfied with the procedure, everything was perfect, I would recommend it to anyone with the same problem.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
units on a scale | 8.22 (1.04) | 7.90 (1.05)
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p = 0.061, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Devices Used
Description: Number of coils and number of vascular plugs used in each procedure
Time Frame: intraoperative
Measure: Mean (Standard Deviation); unit: devices
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
devices | 18.16 (1.33) | 4.06 (0.31)
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Cost of Treatment
Description: Cost of the differential devices used in each treatment procedure, assuming the same cost for the rest of the procedure, other material and hospital stay.
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: US Dollars
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
US Dollars | 3295.05 (240.08) | 4069.79 (138.64)
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Total Intervention Duration
Description: Total time length of the procedure, from puncture to compression (in minutes)
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
minutes | 44.46 (4.09) | 29.02 (5.95)
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

9. Secondary Outcome: Fluoroscopy Time
Description: Total fluoroscopy time, recorded by the equipment (in minutes)
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
minutes | 33.41 (4.68) | 19.52 (6.14)
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

10. Secondary Outcome: Procedure Radiation Dose (DAP)
Description: DAP, dose area product of the intervention, (in mGy*cm^2), recorded by fluoroscopy equipment
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: mGy*cm^2
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
mGy*cm^2 | 354573.00 (105047.76) | 189935.60 (180002.93)
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

11. Secondary Outcome: Procedure Radiation Dose (AK)
Description: AK, total air kerma of the intervention (in mGy), recorded by fluoroscopy equipment
Time Frame: Intraoperative
Measure: Mean (Standard Deviation); unit: mGy
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
mGy | 947.99 (248.45) | 320.66 (134.33)
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Complications
Description: Total number of events during the procedure
Time Frame: intraoperative
Measure: Number; unit: minor events
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
minor events | 11 | 4
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p = 0.0499, Chi-squared

13. Secondary Outcome: Complications
Description: Toral number of events related to the procedure in the follow-up (1 year)
Time Frame: 12 months
Measure: Number; unit: events
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
events | 0 | 0

14. Secondary Outcome: Need for Re-embolization
Description: Scheduled re-embolization due to incomplete occlusion
Time Frame: 12 months
Measure: Number; unit: participants
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Number analyzed (Participants) | 50 | 50
participants
  Re-embolized | 7 | 2
  No | 43 | 48
Statistical Analysis 1: Comparison: Fibered Platinum Coils vs Vascular Plugs; Test type: Superiority or Other; p = 0.095, Fisher Exact

ADVERSE EVENTS:
Time Frame: Intraoperative, 3, 6, and 12 months
Arm/Group | Fibered Platinum Coils | Vascular Plugs
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 11/50 | 5/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fibered Platinum Coils (N=50) | Vascular Plugs (N=50)
Migration of implant or internal device (Vascular disorders) | 3 (3) | 1 (1) — Coil migration to the pulmonary artery. Immediate retrieval during the same intervention. No complications.
Hematoma of neck (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) — Post-puncture hematoma of soft tissues of neck No treatment needed
Extravasation of blood (Vascular disorders) | 6 (6) | 2 (2) — Ovarian vein extravasation assessed during venography. No consequences. No treatment needed.

LIMITATIONS AND CAVEATS:
Analysis of cost dependent on the hospital/region/country. It cannot be extrapolated.

Small number of subjects to compare complication rate of both techniques.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No